CLINICAL TRIAL: NCT03166553
Title: Clinical Trial of Elemene Injection/Elemene Oral Emulsion in Combination With Systematic Chemotherapy Including Oxaliplatin in the First -Line Treatment of Advanced Primary Liver Cancer
Brief Title: Clinical Trial of Elemene in Combination With Oxaliplatinin the Treatment of Advanced Primary Liver Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: BeiJing Yijiayi Medicine Techonoloy Co., Ltd. (Industry)
Collaborators: Dalian Holley Kingkong Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 81YY-ZLLL-16-20
Record Dates: First submitted 2017-05-22; First posted 2017-05-25 (Actual); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Advanced Primary Liver Cancer
MeSH Terms: interventions — elemene; Oxaliplatin

STUDY DESIGN:
Intervention Model Description: One group treated with the Elemene Injection/Elemene Oral Emulusion in Combination with Systematic Chemotherapy including Oxaliplatin , another group treated with Systematic Chemotherapy including Oxaliplatin.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Elemene +Oxaliplatin (Experimental): the group treated with the Elemene Injection/Elemene Oral Emulsion in Combination with Systematic Chemotherapy including Oxaliplatin
  Interventions: Drug: Elemene
- Oxaliplatin (No Intervention): the group treated with Systematic Chemotherapy including Oxaliplatin

INTERVENTIONS:
Drug: Elemene
  Other Names: Oxaliplatin
  Arms: Elemene +Oxaliplatin

SUMMARY:
Clinical Trial of Elemene Injection/Elemene Oral Emulsion in Combination with Systematic Chemotherapy including Oxaliplatin in the First -line treatment of advanced primary liver cancer

DETAILED DESCRIPTION:
Patients with advanced primary liver cancer will be enrolled in the trial , then separated randomly into two group. One group treated with the Elemene Injection/Elemene Oral Emulsion in Combination with Systematic Chemotherapy including Oxaliplatin , another group treated with Systematic Chemotherapy including Oxaliplatin. The purpose of the study is to evaluate the effect and safety of the Elemene Injection/Elemene Oral Emulsion in Combination with Systematic Chemotherapy including Oxaliplatin in the First -line treatment of advanced primary liver cancer

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old，No limit on gender
* Patients who are confirmed Locally advanced or metastatic primary liver cancer in accordance with the clinical diagnostic criteria , or by pathological histology or cytology examination, Patients who are unable to accept surgery,radiofrequency ablation、TACE and local therapy ，orLocal treatment progress failed
* didn't have any systematic treatment including systematic chemotherapy and molecular targeted therapy
* According to RECIST V1.1，1at least has one measurable lesions
* ECOG Score ≤1
* Patients who have primary liver cancer with Child - Pugh liver function grade rating A or better B(score<=7)
* Laboratory inspection basically meets the following requirements：Blood test：a. Hb>=90g/L(without blood transfusion within 14 days), b. ANC>=1.5×10^9/L, c. PLT>=80×10^9/L. Biochemical test：a. ALB>=28g/L(without blood transfusion within 14 days), b. ALT and AST <=5ULN, c. TBIL<=2ULN, d. Cr<=1.5ULN.Blood Coagulation function: PT<=ULN+6seconds
* Life expectancy of at least 3 months
* Subjects join the study voluntarily, sign a consent form, have good compliance, and comply with follow-up

Exclusion Criteria:

* Patients have a adjuvant therapy using Oxaliplatin within 6 months
* Patients have other anti-cancer treatment ， including α-IFN，Arsenious Acid Injection and other Traditional Chinese Medicine Patent Prescription for treating cancer
* Patients blood pressure need to be controled(Systolic blood pressure>150mmHg , Diastolic blood pressure>90mmHg), Congestive heart failure , Unstable angina pectoris , New angina pectoris , and have no Myocardial infarction within 6months
* Patients with severe acute infection and cann't be controled , Chronic suppurative infection , body temperature>=39℃ ， Pleural effusion（medium and large） combined with infection
* Patients with central nervous system metastasis and has symptoms
* In the past or at the same time,patients were diagnosed with other malignant tumor which have not been cured. As for skin basal cell carcinoma and cervical carcinoma in situ,they can be excepted
* Women who is pregnant or during breast feeding and not willing to contraception during the test
* Coagulation dysfunction(PT>16 seconds ， APTT>43 seconds , TT>21 seconds , Fib<2g/L) , With bleeding tendency or the presence of vital organ thrombosis (lung, brain) is receiving thrombolytic or anticoagulant therapy
* With a mental illness, or has a history of drugs abuse
* Patients accepted any experimental drugs in the past 4 weeks
* Other reasons the researchers think not suitable

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-11-28 (Actual); Primary Completion 2019-05-28 (Estimated); Study Completion 2019-11-27 (Estimated)

PRIMARY OUTCOMES:
Objective response rate and/or 1-year survival rate | 1 year
  Objective response rate.The proportion of patients who had a best response rating of complete response and partial response.

SECONDARY OUTCOMES:
Disease control rate(DCR) | 1 year
  Disease control rate.The proportion of patients who had a best response rating of complete response, partial response, or stable disease.
Progression-free survival(PFS) | 1 year
  Progression-free survival.The time of patients from randomization to death caused by the progression of the tumor or any cause
Overall survival(OS) | 3 year
  Overall survival.The time of patient from randomization to death caused by any cause
Quality of Life Questionnaire (QLQ) | 3 year
  Quality of Life Questionnaire Core 30
the rate of incidence of adverse events | 3 year
  NCI CTC AE 4.03

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - 302 Military Hospital of China, Beijing, Beijing Municipality
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Medical University Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiehe University of Science and Technology Affiliate Tongji Hospital, Wuhan, Hubei
  - Jinan Military General Hospital, Jinan, Shandong
  - The Affiliated Hospital of Qindao University, Qindao, Shandong
  - Shanghai Oriental Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No